CLINICAL TRIAL: NCT01053013
Title: An Open-Label Phase 2 Efficacy Trial of the Implantation of Mouse Renal Adenocarcinoma Cell-Containing Agarose-Agarose Macrobeads in the Treatment of Patients With Treatment-Resistant, Metastatic Pancreatic or Colorectal Cancer
Brief Title: Open-Label Phase 2 Efficacy Trial of Cancer Macrobeads in Patients With Treatment-Resistant Pancreatic/Colorectal Cancer
Acronym: Macrobead
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Vital Systems Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0911010739
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable; Pancreatic Adenocarcinoma Metastatic; Colorectal Cancer Metastatic
Keywords: macrobead; biological; mouse cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Macrobead Implantation (Experimental): patients will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at an amount of 8 RENCA macrobeads per kilogram of body weight
  Interventions: Biological: RENCA macrobeads

INTERVENTIONS:
Biological: RENCA macrobeads
  Other Names: mouse renal adenocarcinoma (RENCA) macrobeads; macrobead; cancer macrobead

SUMMARY:
This is a clinical research study of an investigational (FDA BB-IND 10091) treatment for patients with pancreatic cancer (all stages) and advanced colorectal cancer that no longer responds to standard therapies.

The treatment is being evaluated for its effect on tumor growth. It consists of the placement (implantation) of small beads that contain mouse renal adenocarcinoma cells (RENCA macrobeads). The cells in the macrobeads produce substances that have been shown to slow or stop the growth of tumors in experimental animals and veterinary patients. It has been tested in 31 human subjects with different types of cancers in a Phase I safety trial. Phase II studies in patients with colorectal, pancreatic or prostate cancers are in progress.

DETAILED DESCRIPTION:
This is an open-label Phase 2 clinical trial. The study will have a duration of 12 months and involve a potential total of four macrobead implants for each enrolled patient, with the implants being no less than three months apart.

The RENCA macrobeads are implanted intraperitoneally, using laparoscopic surgical procedures. The macrobeads remain permanently within the peritoneal cavity, even if patients withdraw from the study and/or begin new therapy (e.g. chemotherapy). After the formal phase of the trial is completed, subjects will be followed for life.

The intent of this Phase 2 trial is to assess efficacy, safety, and tolerability of RENCA macrobeads. Screening occurs within 28 days prior to first implantation. Enrolled patients are treated with a dose of 8 RENCA macrobeads per kilogram of body weight and observed for a minimum of 3 months prior to the next implantation. A maximum of 4 implantation procedures is possible. Day 0 is the day of implantation.

Prior to the start of the study, the Investigators ensured that the protocol and any attendant documentation were approved, in writing, by the Institutional Review Board. The study was conducted in compliance with the International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use Good Clinical Practice Guidelines (E6 [R1]) for conducting, recording, and reporting studies, as well as for archiving essential documents.

The Investigators, the Medical Monitor of the sponsor, and the Data Safety Monitoring Board were responsible for monitoring safety parameters collected in the study. They, collectively, provided oversight and monitoring of the safety of the participants in the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the pancreas, colon or rectum.
* Radiographic evidence of metastatic cancer of the colon or rectum.
* Pancreatic cancer that is unresectable or already metastatic, or colorectal cancer that has failed available approved treatment modalities.
* For pancreatic cancer patients, prior chemotherapy is not required; for colon and rectal cancer patients must have failed available chemotherapy/targeted regimens. There were no limits to the number of prior chemotherapeutic regimens.
* The patient had evidence of progressive disease defined as at least one of the following:

  1. Progressive measurable disease using conventional solid tumor criteria.
  2. Increasing tumor markers and/or activity on positron emission tomography / standard uptake value (PET/SUV) measurement.
* All clinically significant toxic effects (excluding alopecia) of prior surgery, radiotherapy, or hormonal therapy were resolved to ≤ Grade 1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0 (NCI CTCAE v.3.0) with the exception of neuropathy, which was resolved to ≤ Grade 2.
* Performance status (ECOG PS) 0-2.
* Adequate hematologic function, minimum requirements:

  1. absolute neutrophil count (ANC) ≥ 1500/mL
  2. hemoglobin ≥ 9 g/dL
  3. platelets ≥ 100,000/mL
* Adequate hepatic function, defined as follows:

  1. bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  2. aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times the ULN, or ≤ 5 times the ULN if liver metastases are present
* Adequate renal function, defined as serum creatinine ≤ 2.0 mg/dL.
* Adequate coagulation function, defined as follows:

  1. an international normalized ratio (INR) ≤ 1.5
  2. a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN, unless on anti-coagulant therapy
  3. patients receiving full-dose anticoagulation therapy were eligible provided they met all other criteria, were on a stable dose or anticoagulant therapy or low molecular weight heparin (and if on warfarin had a therapeutic INR between 2-3)
* Life expectancy of at least 6 weeks.
* For females of childbearing potential, a negative pregnancy test.
* Agrees to contraceptive use (barrier method) while on study, if sexually active.
* Provided signed informed consent.

Exclusion Criteria:

* Any condition presenting an unacceptably high anesthetic or surgical risk, based on current anesthesia/general surgery standards.
* Positive test for HIV, hepatitis B, C, or E.
* Cognitive impairment such as to preclude informed consent.
* Hypersensitivity reaction that, in the opinion of the investigators posed an increased risk of an allergy to the macrobeads, particularly any known allergy to murine antigens or body tissues.
* Surgical treatment or chemotherapy within three weeks of scheduled macrobead implantation or within four weeks of bevacizumab (or similar drugs), or radiation therapy within four weeks of scheduled macrobead implantation.
* Investigational medication(s)/therapies for respective tumor within one month of baseline evaluation.
* Inadequate hematologic function, defined as follows:

  1. ANC < 1500/mL
  2. hemoglobin < 9 g/dL
  3. platelets < 100,000/mL
* Inadequate hepatic function, defined as follows:

  1. bilirubin > 1.5 times the ULN
  2. AST and ALT > 3 times the ULN or > 5 times the ULN, if liver metastases present
* Inadequate renal function, defined as serum creatinine > 2.0 mg/dL.
* Inadequate coagulation function, defined as follows:

  1. INR > 1.5
  2. PTT > 5 seconds (unless on anti-coagulant therapy)
* Hepatic blood flow abnormalities, portal vein hypertension and thrombosis, and/or large-volume ascites.
* Concurrent cancer of any other type except skin cancer (excluding melanoma).
* Ongoing or active infection, congestive heart failure, unstable angina, serious cardiac arrhythmias, psychiatric illness, difficult social situations not permitting reliable participation, active bleeding.
* As a result of the medical history, examination, or blood testing, the investigator considers the patient unfit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-04-15 (Actual); Primary Completion 2016-04-16 (Actual); Study Completion 2016-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fahey, III., MD, Principal Investigator — Weill Cornell Medical Center / New York-Presbyterian Hospital
Locations (1):
- Weill Cornell Medical Center / The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Three-dimensional culture of mouse renal carcinoma cells in agarose macrobeads selects for a subpopulation of cells with cancer stem cell or cancer progenitor properties. Cancer Res. 2011 Feb 1;71(3):716-24. doi: 10.1158/0008-5472.CAN-10-2254. Epub 2011 Jan 24. PMID 21266363
- [Background] Smith BH, Gazda LS, Conn BL, Jain K, Asina S, Levine DM, Parker TS, Laramore MA, Martis PC, Vinerean HV, David EM, Qiu S, North AJ, Couto CG, Post GS, Waters DJ, Cordon-Cardo C, Hall RD, Gordon BR, Diehl CH, Stenzel KH, Rubin AL. Hydrophilic agarose macrobead cultures select for outgrowth of carcinoma cell populations that can restrict tumor growth. Cancer Res. 2011 Feb 1;71(3):725-35. doi: 10.1158/0008-5472.CAN-10-2258. Epub 2011 Jan 24. PMID 21266362
- [Background] Smith BH, Gazda LS, Fahey TJ, Nazarian A, Laramore MA, Martis P, Andrada ZP, Thomas J, Parikh T, Sureshbabu S, Berman N, Ocean AJ, Hall RD, Wolf DJ. Clinical laboratory and imaging evidence for effectiveness of agarose-agarose macrobeads containing stem-like cells derived from a mouse renal adenocarcinoma cell population (RMBs) in treatment-resistant, advanced metastatic colorectal cancer: Evaluation of a biological-systems approach to cancer therapy (U.S. FDA IND-BB 10091; NCT 02046174, NCT 01053013). Chin J Cancer Res. 2018 Feb;30(1):72-83. doi: 10.21147/j.issn.1000-9604.2018.01.08. PMID 29545721
- [Background] Gazda LS, Martis PC, Laramore MA, Bautista MA, Dudley A, Vinerean HV, Smith BH. Treatment of agarose-agarose RENCA macrobeads with docetaxel selects for OCT4(+) cells with tumor-initiating capability. Cancer Biol Ther. 2013 Dec;14(12):1147-57. doi: 10.4161/cbt.26455. Epub 2013 Sep 12. PMID 24025409
- [Background] Martis PC, Dudley AT, Bemrose MA, Gazda HL, Smith BH, Gazda LS. MEF2 plays a significant role in the tumor inhibitory mechanism of encapsulated RENCA cells via EGF receptor signaling in target tumor cells. BMC Cancer. 2018 Dec 4;18(1):1217. doi: 10.1186/s12885-018-5128-5. PMID 30514247
- [Background] Smith BH, Parikh T, Andrada ZP, Fahey TJ, Berman N, Wiles M, Nazarian A, Thomas J, Arreglado A, Akahoho E, Wolf DJ, Levine DM, Parker TS, Gazda LS, Ocean AJ. First-in-Human Phase 1 Trial of Agarose Beads Containing Murine RENCA Cells in Advanced Solid Tumors. Cancer Growth Metastasis. 2016 Aug 2;9:9-20. doi: 10.4137/CGM.S39442. eCollection 2016. PMID 27499645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral between April 2010 and February 2016. The first participant was implanted on April 15, 2010 (pancreatic) and May 14, 2010 (mCRC). The last implantation was on March 4, 2016 (pancreatic) and October 18, 2013 (mCRC).
Pre-assignment Details: 90 participants provided informed consent to participate in the study (Pancreatic cancer n=34; mCRC n=46). Of these, 24 pancreatic cancer patients and 34 mCRC patients were enrolled in the study. The 22 patients who were not enrolled into the study, after providing consent, had failed the respective eligibility criteria (n=19) or decided not to enroll in the study (n=3).
Groups:
- Pancreatic Cancer: Pancreatic cancer patients will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
  RENCA Macrobeads.
- Metastatic Colorectal Cancer: Metastatic colorectal cancer (mCRC) patients who will undergo up to 4 implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
  RENCA macrobeads
Period: Overall Study
Arm/Group | Pancreatic Cancer | Metastatic Colorectal Cancer
Started | 24 | 34
Completed | 24 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pancreatic Cancer | Metastatic Colorectal Cancer | Total
Number analyzed (Participants) | 24 | 34 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.25 (12.37) | 58.00 (10.11) | 58.93 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 16 | 11 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 27 | 49
  Black | 1 | 4 | 5
  Hispanic | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native American | 0 | 0 | 0
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival - Based on Most Recent Scan
Description: The primary efficacy outcome is post-implantation all-cause mortality, where time to death is defined as the time from the most recent scan prior to first implantation (time of origin, To) to death from any cause.
Time Frame: From date of the most recent scan (disease progression) prior to the first macrobead implantation; assessed up to 32 months.
Population: Participants who received at least one RENCA macrobead implant.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pancreatic Cancer | Metastatic Colorectal Cancer
Number analyzed (Participants) | 24 | 34
months | 4.66 [2.43 to 5.74] | 7.7 [6.1 to 12.2]

2. Secondary Outcome: Overall Survival - Based on 1st Implant
Description: The secondary efficacy objective was to evaluate overall survival calculated using the time from first RENCA macrobead implantation to death from any cause.
Time Frame: From date of the first RENCA macrobead implant; assessed up to 32 months.
Population: Participants who received at least one RENCA macrobead implant.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pancreatic Cancer | Metastatic Colorectal Cancer
Number analyzed (Participants) | 24 | 34
months | 4.3 [2.03 to 5.18] | 7.3 [5.4 to 11.4]

3. Other Pre Specified Outcome: Necrosis Comparison of Tumors Using PET-CT Scan
Description: Tumors were assessed by positron emission tomography (PET)-CT scan at baseline and day 90 following the first RENCA macrobead implantation. The use of [13]F-fluorodeoxyglucose (FDG) uptake for the detection of lesions >1 cm in diameter allowed evaluation of metabolic activity. Decreases in FDG uptake were indicative of metabolic suppression of the tumor. The use of PET-CT scanning indicated anatomical localization, approximate size/volume of primary tumor and metastatic lesion(s), and assessment of metabolic activity of the tumor (as an indicator of metabolic health and necrosis).
  Disease state is reported as a function of Tumor measurement divided by SUVmax. Changes were assessed between day 90 post RENCA macrobead implant and baseline values. Patients with no change = stable; patients with decreased values = decreased/necrosis, and patients with increased values = increased.
Time Frame: Baseline vs. Day 90 post-Implant 1
Population: mCRC participants who had received at least one macrobead implant and for whom baseline PET-CT scan and day 90 post-Implant 1 PET-CT scan data were available. n=26 subjects; 77 lesions evaluated. No formal analysis was performed on the pancreatic cancer cohort as a meaningful analysis was limited based on the small group size with baseline and day 90 scans.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- Stable: mCRC participants with stable disease based on imaging results [Tumor measurements/SUV max].
- Decreased/Necrosis: mCRC participants with decreased/necrosis observed based on imaging results [Tumor measurements/SUV max].
- Increased: mCRC participants with increased SUVmax, tumor measurement based on imaging results.
Arm/Group | Stable | Decreased/Necrosis | Increased
Number analyzed (Participants) | 26 | 26 | 26
Number analyzed (lesions) | 87 | 87 | 87
lesions | 15 | 42 | 30

4. Other Pre Specified Outcome: Tumor Marker Response of mCRC Participants
Description: Tumor markers included serum carcinoembryonic antigen (CEA) and cancer antigen 19-9 (CA 19-9), and were assessed on all participants with mCRC at baseline and at subsequent evaluation points to further assess tumor response to RENCA macrobead implantation. A tumor marker response was defined as a greater than or equal to 20% decrease in one or both of CEA or CA 19-9.
Time Frame: Change from baseline up to and including day 30 post-Implant 1
Population: Participants with mCRC receiving at least one RENCA macrobead implantation.
Measure: Count of Participants; unit: Participants
Groups:
- mCRC: CEA Only: Participants with mCRC whose tumor marker response was greater than or equal to 20% decrease from baseline in CEA only [up to and including day 90 after the first implant).
- mCRC CA 19-9 Only: Participants with mCRC whose tumor marker response was greater than or equal to 20% decrease from baseline in CA 19-9 only [up to and including day 90 after the first implant).
- mCRC: Both CEA and CA 19-9: Participants with mCRC whose tumor marker response was greater than or equal to 20% decrease from baseline in both CEA and CA 19-9 [up to and including day 90 after the first implant).
- mCRC: Non-responder: Participants with mCRC whose tumor marker response (serum level of CEA and/or CA 19-9) did not decrease by greater than or equal to 20% of baseline value.
Arm/Group | mCRC: CEA Only | mCRC CA 19-9 Only | mCRC: Both CEA and CA 19-9 | mCRC: Non-responder
Number analyzed (Participants) | 34 | 34 | 34 | 34
Participants | 7 | 3 | 15 | 9

5. Other Pre Specified Outcome: Tumor Marker Response of Pancreatic Cancer Participants
Description: Tumor markers included serum carcinoembryonic antigen (CEA) and cancer antigen 19-9 (CA 19-9), and were assessed on all participants with pancreatic cancer at baseline and at subsequent evaluation points to further assess tumor response to RENCA macrobead implantation. A tumor marker response was defined as a greater than or equal to 20% decrease in one or both of CEA or CA 19-9.
Time Frame: Change from baseline up to and including day 30 post-Implant 1.
Population: Participants with pancreatic cancer receiving at least one RENCA macrobead implantation.
Measure: Count of Participants; unit: Participants
Groups:
- Pancreatic Cancer: CEA Only: Participants with pancreatic cancer whose tumor marker response was greater than or equal to 20% decrease from baseline in CEA only [up to and including day 90 after the first implant).
- Pancreatic Cancer: CA 19-9 Only: Participants with pancreatic cancer whose tumor marker response was greater than or equal to 20% decrease from baseline in CA 19-9 only [up to and including day 90 after the first implant).
- Pancreatic Cancer: Both CEA and CA 19-9: Participants with pancreatic cancer whose tumor marker response was greater than or equal to 20% decrease from baseline in both CEA and CA 19-9 [up to and including day 90 after the first implant).
- Pancreatic Cancer: Non-responder: Participants with pancreatic cancer whose tumor marker response (serum level of CEA and/or CA 19-9) did not decrease by greater than or equal to 20% of baseline value.
Arm/Group | Pancreatic Cancer: CEA Only | Pancreatic Cancer: CA 19-9 Only | Pancreatic Cancer: Both CEA and CA 19-9 | Pancreatic Cancer: Non-responder
Number analyzed (Participants) | 24 | 24 | 24 | 24
Participants | 3 | 1 | 6 | 14

6. Other Pre Specified Outcome: C-reactive Protein Levels in mCRC Participants
Description: C-reactive protein (CRP) is one of three inflammatory markers assessed during this study. CRP levels were assessed as a marker of systemic inflammatory processes.
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: Implant 1 (Days 0-60): Participants with mCRC who had received at least 1 RENCA macrobead implantation and were screened as indicated; Implant 2 (Days 0-60): Participants with mCRC who had received at least 2 RENCA macrobead implantations and were screened as indicated. In some cases, participants may not have had all assessments conducted as scheduled. In those incidents, the number of participants analyzed has been adjusted to include only those participants for which data was available.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Implant 1: Day 0: CRP levels at baseline, prior to first implantation.
- Implant 1: Day 14: CRP levels at day 14 after first implantation.
- Implant 1: Day 30: CRP levels at day 30 after first implantation.
- Implant 1: Day 60: CRP levels at day 60 after first implantation.
- Implant 2: Day 0: CRP levels at day 0 of second implantation (day 90 following first implantation).
- Implant 2: Day 14: CRP levels at day 14 after second implantation.
- Implant 2: Day 30: CRP levels at day 30 after second implantation.
- Implant 2: Day 60: CRP levels at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 34 | 34 | 30 | 13 | 12 | 13 | 11
mg/dL | 3.1 (4.2) | 19.3 (8.1) | 8.9 (5.9) | 6.7 (6.9) | 10.2 (23.6) | 23.5 (50.8) | 11.4 (8.3) | 5.5 (4.1)

7. Other Pre Specified Outcome: C-Reactive Protein Levels in Pancreatic Cancer Participants
Description: as for outcome 6
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: Implant 1 (Days 0-60): Pancreatic cancer participants who had received at least 1 implant and were screened as indicated; Implant 2 (Days 0-60): Pancreatic cancer participants who had received at least 2 RENCA macrobead implantations and were screened as indicated. In some cases, participants may not have had all assessments conducted as scheduled. In those incidents, the number of participants analyzed has been adjusted to include only those participants for which data was available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 21 | 20 | 15 | 3 | 3 | 3 | 1
mg/dL | 1.7 (2.0) | 30.7 (46.7) | 13.8 (22.9) | 6.7 (11.6) | 1.4 (1.3) | 3.1 (1.7) | 89.8 (148.4) | 7.52

8. Other Pre Specified Outcome: Erythrocyte Sedimentation Rate in mCRC Participants
Description: Erythrocyte sedimentation rate (ESR) is one of three inflammatory markers assessed during this study. ESR was assessed as a marker of systemic inflammatory processes.
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm/hr
Groups:
- Implant 1: Day 0: ESR at baseline, prior to first implantation.
- Implant 1: Day 14: ESR at day 14 after first implantation.
- Implant 1: Day 30: ESR at day 30 after first implantation.
- Implant 1: Day 60: ESR at day 60 after first implantation.
- Implant 2: Day 0: ESR at day 0 of second implantation (day 90 following first implantation).
- Implant 2: Day 14: ESR at day 14 after second implantation.
- Implant 2: Day 30: ESR at day 30 after second implantation.
- Implant 2: Day 60: ESR at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 34 | 32 | 30 | 13 | 10 | 12 | 10
mm/hr | 44.9 (30.9) | 92.7 (31.4) | 85.8 (37.3) | 68.1 (39.6) | 53.5 (16.1) | 93.3 (27.7) | 92.7 (23.1) | 74.9 (28.8)

9. Other Pre Specified Outcome: Erythrocyte Sedimentation Rate in Pancreatic Cancer Participants
Description: as for outcome 8
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 23 | 18 | 18 | 11 | 3 | 2 | 1 | 0
mm/hr | 33 (24.6) | 51.9 (31.3) | 49.2 (12.9) | 78.6 (13.8) | 83.3 (5.8) | 90.0 (14.1) | 80.0 |

10. Other Pre Specified Outcome: Cancer Antigen 125 Levels in mCRC Participants
Description: Cancer Antigen 125 (CA 125) is one of three inflammatory markers assessed during this study. CA 125 was used to monitor more localized intra-abdominal/peritoneal inflammatory processes related to the placement of the RENCA macrobeads or, in some cases, the intraperitoneal spread of tumor.
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/mL
Groups:
- Implant 1: Day 0: CA 125 levels at baseline, prior to first implantation.
- Implant 1: Day 14: CA 125 levels at day 14 after first implantation.
- Implant 1: Day 30: CA 125 levels at day 30 after first implantation.
- Implant 1: Day 60: CA 125 levels at day 60 after first implantation.
- Implant 2: Day 0: CA 125 levels at day 0 of second implantation (day 90 following first implantation).
- Implant 2: Day 14: CA 125 levels at day 14 after second implantation.
- Implant 2: Day 30: CA 125 levels at day 30 after second implantation.
- Implant 2: Day 60: CA 125 levels at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 33 | 34 | 30 | 13 | 12 | 13 | 11
U/mL | 43.5 (76.65) | 95.5 (73.5) | 83.7 (86.6) | 67.6 (106.1) | 39.2 (49.1) | 63.7 (29.1) | 48.7 (31.4) | 38.0 (31.9)

11. Other Pre Specified Outcome: Cancer Antigen 125 Levels in Pancreatic Cancer Participants
Description: as for outcome 10
Time Frame: Day 0, 14, 30, 60 post-Implant 1 and Day 0, 14, 30, 60 post-Implant 2 (when applicable).
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 23 | 21 | 20 | 15 | 3 | 2 | 2 | 1
U/mL | 147.9 (278.6) | 300.7 (410.6) | 409.4 (607.0) | 291.7 (289.2) | 49.7 (30.1) | 88.5 (7.8) | 117.0 (46.7) | 57.0

12. Other Pre Specified Outcome: Performance Status (ECOG Score) of mCRC Participants
Description: The Eastern Cooperative Oncology Group (ECOG) performance scale is a 5-point scale, where 0 denotes perfect health and 5 is death. It is used by clinicians to assess disease progression and how the disease is affecting the daily living abilities of the patient. The ECOG Performance Status scores are defined as follows:
  0: Fully active, able to carry on all pre-disease activities without restriction.
  1. Restricted in physical strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g. light house work, office work).
  2. Ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair 50% or more of waking hours.
  4. Completely disabled, cannot carry on any self-care, totally confined to bed or chair.
  5. Death
Time Frame: Baseline; Day 14, 30, 60 post-Implant; Day 14, 30, 60 post-Implant 2
Population: Implant (day 0 to day 60): Participants with mCRC who received at least one RENCA macrobead implantation; Implant 2 (day 0 to day 60): Participants who received at least two RENCA macrobead implantations.
Measure: Count of Participants; unit: Participants
Groups:
- Implant 1: Day 0: ECOG score at pre-screening for first implantation.
- Implant 1: Day 14: ECOG score at day 14 after first implantation.
- Implant 1: Day 30: ECOG score at day 30 after first implantation.
- Implant 1: Day 60: ECOG score at day 60 after first implantation.
- Implant 2: Day 0: ECOG score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: ECOG score at day 14 after second implantation.
- Implant 2: Day 30: ECOG score at day 30 after second implantation.
- Implant 2: Day 60: ECOG score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 28 | 25 | 24 | 24 | 12 | 6 | 9 | 9
Participants
  ECOG Score 0 | 13 | 4 | 3 | 4 | 5 | 0 | 2 | 1
  ECOG Score 1 | 15 | 15 | 16 | 10 | 5 | 3 | 4 | 5
  ECOG Score 2 | 0 | 5 | 3 | 6 | 2 | 3 | 3 | 2
  ECOG Score 3 | 0 | 1 | 2 | 4 | 0 | 0 | 0 | 1
  ECOG Score 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ECOG Score 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Performance Status (ECOG Score) of Pancreatic Cancer Participants
Description: as for outcome 12
Time Frame: Baseline; Day 14, 30, 60 post-Implant; Day 14, 30, 60 post-Implant 2
Population: Implant 1 (Days 0-60): Pancreatic cancer participants who had received at least 1 macrobead implantation and were screened as indicated; Implant 2 (Days 0-60): Pancreatic cancer participants who had received at least 2 macrobead implantations and were screened as indicated. In some cases, participants may not have had all assessments conducted as scheduled. In those incidents, the number of participants analyzed has been adjusted to include only those participants for which data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 23 | 20 | 16 | 12 | 3 | 2 | 2 | 0
Participants
  ECOG Score 0 | 11 | 1 | 3 | 4 | 1 | 1 | 0 |
  ECOG Score 1 | 7 | 11 | 8 | 4 | 1 | 1 | 2 |
  ECOG Score 2 | 5 | 7 | 5 | 2 | 1 | 0 | 0 |
  ECOG Score 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0 |
  ECOG Score 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  ECOG Score 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

14. Other Pre Specified Outcome: Activities of Daily Living (KPS Score) of mCRC Participants
Description: Karnofsky Performance Status (KPS) is a self-rated scale that measures the participant's ability to perform daily functions, ranging from 0 ("dead") to 100 ("normal, no complaints, no evidence of disease). Karnofsky scores are defined as follows:
  100: Normal; no complaints; no evidence of disease 90: Able to carry on normal activity with effort, minor sign or symptoms of disease 80: Normal activity with effort; some sign or symptoms of disease 70: Cares for self; unable to carry on normal activity or do active work 60: Requires occasional assistance, but is able to care for most personal needs 50: Requires considerable assistance and frequent medical care 40: Disabled; requires special care and assistance 30: Severely disabled; hospitalization is indicated, although death is not imminent 20: Very sick; hospitalization/active support treatment is necessary 10: Moribund; fatal processes progressively worsening 0: Dead
Time Frame: Baseline; Day 14, 30, 60 Post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: KPS score at pre-screening for first implantation.
- Implant 1: Day 14: KPS score at day 14 after first implantation.
- Implant 1: Day 30: KPS score at day 30 after first implantation.
- Implant 1: Day 60: KPS score at day 60 after first implantation.
- Implant 2: Day 0: KPS score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: KPS score at day 14 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 32 | 26 | 27 | 28 | 13 | 8 | 11 | 10
score on a scale | 90.0 (7.2) | 81.2 (11.8) | 80.4 (11.6) | 74.1 (16.6) | 84.2 (9.1) | 76.3 (11.9) | 82.7 (9.1) | 76.0 (16.5)

15. Other Pre Specified Outcome: Activities of Daily Living (KPS Score) for Pancreatic Cancer Participants
Description: as for outcome 14
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 2: Day 30: KPS score at day 30 after second implantation.
- Implant 2: Day 60: KPS score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 19 | 14 | 11 | 3 | 2 | 1 | 0
score on a scale | 87.9 (9.3) | 79.5 (9.7) | 78.6 (12.9) | 78.6 (13.8) | 83.3 (5.8) | 90.0 (14.1) | 80.0 |

16. Other Pre Specified Outcome: Global Health Status of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales, three symptom scales, a global health status score, and six single items.
  The Global Health Status is assessed from 2 of the 30 questions (Question 29 and 30), whose response score ranges on a 7 point scale. The score for physical function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor) and the maximum value is 100 (best outcome, excellent). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: Global health status score at pre-screening for first implantation.
- Implant 1: Day 14: Global health status score at day 14 after first implantation.
- Implant 1: Day 30: Global health status score at day 30 after first implantation.
- Implant 1: Day 60: Global health status score at day 60 after first implantation.
- Implant 2: Day 0: Global health status score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: Global health status score at day 14 after second implantation.
- Implant 2: Day 30: Global health status score at day 30 after second implantation.
- Implant 2: Day 60: Global health status score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 32 | 25 | 26 | 26 | 13 | 7 | 10 | 9
score on a scale | 94.0 (8.4) | 78.8 (15.9) | 80.6 (17.3) | 75.1 (25.9) | 86.0 (11.4) | 78.6 (9.6) | 86.7 (9.5) | 83.3 (16.7)

17. Other Pre Specified Outcome: Global Health Status of Pancreatic Cancer Participants
Description: as for outcome 16
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 16 | 14 | 10 | 3 | 1 | 1 | 0
score on a scale | 90.1 (10.8) | 75.2 (18.8) | 77.8 (15.9) | 72.3 (24.3) | 84.2 (4.6) | 26.5 | 25.6 |

18. Other Pre Specified Outcome: Physical Function of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including physical function), three symptom scales, a global health status score, and six single items.
  Physical Function is assessed from 5 of the 30 questions (Questions 1-5), whose response score ranges on a 4 point scale. The score for physical function is calculated based on the average score from these 5 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: Implant 1 (Day 0 to Day 60): Participants with mCRC who had received at least 1 RENCA macrobead implantation; Implant 2 (Day 0 to Day 60): Participants with mCRC who had received at least 2 RENCA macrobead implantations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Physical functioning score at pre-screening for first implantation.
- Implant 1: Day 30: EORTC/Physical functioning score at day 30 after first implantation.
- Implant 1: Day 60: EORTC/Physical functioning score at day 60 after first implantation.
- Implant 2: Day 0: EORTC/Physical functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 30: EORTC/Physical functioning score at day 30 after second implantation.
- Implant 2: Day 60: EORTC/Physical functioning score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 32 | 30 | 28 | 13 | 10 | 9
score on a scale | 86.9 (16.2) | 69.8 (26.9) | 66.9 (28.4) | 78.5 (16.8) | 66.7 (25.5) | 63.7 (35.0)

19. Other Pre Specified Outcome: Physical Function of Pancreatic Cancer Participants
Description: as for outcome 18
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: Implant 1 (Day 0 to Day 60): Pancreatic cancer participants who had received at least 1 macrobead implantation; Implant 2 (Day 0 to Day 60): Pancreatic cancer participants who had received at least 2 macrobead implantations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 19 | 13 | 3 | 2 | 0
score on a scale | 81.1 (20.6) | 62.5 (28.5) | 64.1 (33.7) | 91.1 (10.2) | 76.7 (23.6) |

20. Other Pre Specified Outcome: Role Function of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including role function), three symptom scales, a global health status score, and six single items.
  Role Function is assessed from 2 of the 30 questions (Questions 6 and 7), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Role functioning score at pre-screening for first implantation.
- Implant 1: Day 30: EORTC/Role functioning score at day 30 after first implantation.
- Implant 1: Day 60: EORTC/Role functioning score at day 60 after first implantation.
- Implant 2: Day 0: EORTC/Role functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 30: EORTC/Role functioning score at day 30 after second implantation.
- Implant 2: Day 60: EORTC/Role functioning score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 32 | 30 | 28 | 13 | 10 | 9
score on a scale | 85.9 (17.5) | 58.3 (29.3) | 56.0 (36.9) | 75.6 (32.4) | 55.0 (36.9) | 51.9 (32.8)

21. Other Pre Specified Outcome: Role Function of Pancreatic Cancer Participants
Description: as for outcome 20
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: Implant 1 (Day 0 to Day 60): Participants with pancreatic cancer who had received at least 1 RENCA macrobead implantation; Implant 2 (Day 0 to Day 60): Participants with pancreatic cancer who had received at least 2 RENCA macrobead implantations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 19 | 13 | 3 | 2 | 0
score on a scale | 80.6 (27.2) | 58.5 (32.3) | 52.6 (36.5) | 83.3 (16.7) | 50.0 (23.6) |

22. Other Pre Specified Outcome: Emotional Function of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including emotional function), three symptom scales, a global health status score, and six single items.
  Emotional Function is assessed from 4 of the 30 questions (Questions 21-24), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 4 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Emotional functioning score at pre-screening for first implantation.
- Implant 1: Day 30: EORTC/Emotional functioning score at day 30 after first implantation.
- Implant 2: Day 0: EORTC/Emotional functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 30: EORTC/Emotional functioning score at day 30 after second implantation.
- Implant 2: Day 60: EORTC/Emotional functioning score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 30 | 27 | 13 | 10 | 9
score on a scale | 83.3 (18.5) | 78.1 (18.4) | 74.3 (22.2) | 84.0 (16.8) | 75.8 (21.3) | 75.9 (17.4)

23. Other Pre Specified Outcome: Emotional Function of Pancreatic Cancer Participants
Description: as for outcome 22
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 18 | 13 | 3 | 2 | 0
score on a scale | 82.3 (20.3) | 70.4 (30.9) | 69.2 (32.9) | 91.7 (14.4) | 83.3 (11.8) |

24. Other Pre Specified Outcome: Cognitive Function of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including cognitive function), three symptom scales, a global health status score, and six single items.
  Cognitive Function is assessed from 2 of the 30 questions (Question 20 and 25), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Cognitive functioning score at pre-screening for first implantation.
- Implant 1: Day 30: EORTC/Cognitive functioning score at day 30 after first implantation.
- Implant 1: Day 60: EORTC/Cognitive functioning score at day 60 after first implantation.
- Implant 2: Day 0: EORTC/Cognitive functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 30: EORTC/Cognitive functioning score at day 30 after second implantation.
- Implant 2: Day 60: EORTC/Cognitive functioning score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 30 | 27 | 13 | 10 | 9
score on a scale | 86.9 (18.5) | 84.4 (19.0) | 82.1 (25.3) | 79.5 (22.7) | 71.7 (24.9) | 72.2 (30.0)

25. Other Pre Specified Outcome: Cognitive Function of Pancreatic Cancer Participants
Description: as for outcome 24
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 18 | 13 | 13 | 10 | 9
score on a scale | 87.5 (18.6) | 72.2 (39.2) | 73.1 (36.3) | 79.5 (22.7) | 71.7 (24.9) | 72.2 (30.0)

26. Other Pre Specified Outcome: Social Function of mCRC Participants
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3.0) consists of 30 questions which pertain to: five functional scales (including social function), three symptom scales, a global health status score, and six single items.
  Social Function is assessed from 2 of the 30 questions (Question 26 and 27), whose response score ranges on a 4 point scale. The score for role function is calculated based on the average score from these 2 questions. A linear transformation is used to standardize these responses. Using this linear transformation, the minimum value is 0 (worst outcome, poor functionality) and the maximum value is 100 (best outcome, better functionality). Therefore, increasing values indicate better outcome and decreasing values indicate worse outcome.
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: EORTC/Social functioning score at pre-screening for first implantation.
- Implant 1: Day 30: EORTC/Social functioning score at day 30 after first implantation.
- Implant 1: Day 60: EORTC/Social functioning score at day 60 after first implantation.
- Implant 2: Day 0: EORTC/Social functioning score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 30: EORTC/Social functioning score at day 30 after second implantation.
- Implant 2: Day 60: EORTC/Social functioning score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 33 | 30 | 27 | 13 | 10 | 9
score on a scale | 82.8 (21.8) | 67.2 (30.5) | 59.9 (36.5) | 70.5 (27.3) | 60.0 (27.4) | 53.7 (35.1)

27. Other Pre Specified Outcome: Social Function of Pancreatic Cancer Participants
Description: as for outcome 26
Time Frame: Baseline; Day 30, 60 post-Implant 1; Day 30, 60 post-Implant 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 24 | 17 | 13 | 3 | 2 | 0
score on a scale | 76.4 (31.1) | 58.8 (30.1) | 61.5 (33.6) | 77.8 (19.2) | 50.0 (0.0) |

28. Other Pre Specified Outcome: Pain Assessment of mCRC Participants
Description: Participants were asked to rate their pain on a discrete scale (from 0 = "no pain" to 10 "worst pain imaginable, unbearable"). The worst pain at each time point was used in the analysis.
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implant 1: Day 0: Pain assessment score at pre-screening for first implantation.
- Implant 1: Day 14: Pain assessment score at day 14 after first implantation.
- Implant 1: Day 30: Pain assessment score at day 30 after first implantation.
- Implant 1: Day 60: Pain assessment score at day 60 after first implantation.
- Implant 2: Day 0: Pain assessment score at pre-screening for second implantation (day 90 following first implantation).
- Implant 2: Day 14: Pain assessment score at day 14 after second implantation.
- Implant 2: Day 30: EORTC/Pain assessment score at day 30 after second implantation.
- Implant 2: Day 60: Pain assessment score at day 60 after second implantation.
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 28 | 24 | 26 | 24 | 13 | 7 | 11 | 10
score on a scale | 1.7 (2.7) | 3.3 (3.0) | 2.5 (2.4) | 3.8 (2.7) | 2.2 (2.8) | 5.4 (2.2) | 4.2 (3.0) | 4.2 (3.6)

29. Other Pre Specified Outcome: Pain Assessment of Pancreatic Cancer Participants
Description: as for outcome 28
Time Frame: Baseline; Day 14, 30, 60 post-Implant 1; Day 14, 30, 60 post-Implant 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implant 1: Day 0 | Implant 1: Day 14 | Implant 1: Day 30 | Implant 1: Day 60 | Implant 2: Day 0 | Implant 2: Day 14 | Implant 2: Day 30 | Implant 2: Day 60
Number analyzed (Participants) | 23 | 17 | 15 | 10 | 3 | 1 | 2 | 0
score on a scale | 1.5 (2.1) | 2.3 (3.2) | 2.9 (2.5) | 3.9 (2.4) | 5.5 (3.0) | 4.0 | 3.7 (1.8) |

30. Secondary Outcome: Overall Survival - Based on Stage IV Disease Diagnosis
Description: The secondary efficacy objective was to evaluate overall survival calculated using the time from Stage IV disease diagnosis to death from any cause.
Time Frame: From date of Stage IV disease diagnosis up to 126 months; up to 32 months from first RENCA macrobead implant.
Population: Participants who received at least one RENCA macrobead implant.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pancreatic Cancer | Metastatic Colorectal Cancer
Number analyzed (Participants) | 24 | 34
months | 15.7 [11.97 to 18.89] | 32.1 [27.2 to 43.2]

ADVERSE EVENTS:
Time Frame: From date of first macrobead implantation; assessed up to 32 months.
Description: The NCI CTCAE was used to standardize the terminology and grade the severity of reported adverse events. The Principal and Sub-Investigators, and Attending Physicians, were responsible for monitoring adverse events and the safety of all participants. The Data Safety Monitoring Board, independently and in collaboration with the PIs, monitored and reviewed all safety findings, including study status, serious adverse events, AEs > Grade 2, laboratory values of special interest and subject deaths.
Groups:
- Metastatic Colorectal Cancer (mCRC) Participants: Metastatic colorectal cancer (mCRC) patients who underwent at least 1 (and up to 4) implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
- Pancreatic Cancer Participants: Pancreatic cancer patients who underwent at least 1 (and up to 3) implantations of RENCA macrobeads (no less than 3 months apart), at a dosage level of 8 RENCA macrobeads per kilogram of body weight.
Arm/Group | Metastatic Colorectal Cancer (mCRC) Participants | Pancreatic Cancer Participants
All-Cause Mortality (participants affected / at risk) | 34/34 | 24/24
Serious Adverse Events (participants affected / at risk) | 31/34 | 20/24
Other Adverse Events (participants affected / at risk) | 34/34 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Colorectal Cancer (mCRC) Participants (N=34) | Pancreatic Cancer Participants (N=24)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Adominal pain (Gastrointestinal disorders) | 2 | 5
Ascites (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 24 | 13
Asthenia (General disorders) | 2 | 0
Hernia (General disorders) | 2 | 0
Pain (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Abdominal ascites (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac enzymes increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm of paraurethral glands (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Inferior vena caval occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metastatic Colorectal Cancer (mCRC) Participants (N=34) | Pancreatic Cancer Participants (N=24)
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 9 | 4
Abdominal pain (Gastrointestinal disorders) | 23 | 11
Constipation (Gastrointestinal disorders) | 15 | 14
Nausea (Gastrointestinal disorders) | 19 | 10
Abdominal distension (Gastrointestinal disorders) | 12 | 9
Vomiting (Gastrointestinal disorders) | 14 | 6
Diarroea (Gastrointestinal disorders) | 11 | 9
Ascites (Gastrointestinal disorders) | 3 | 6
Flatulance (Gastrointestinal disorders) | 4 | 4
Abdominal pain discomfort (Gastrointestinal disorders) | 5 | 1
Abdominal pain lower (Gastrointestinal disorders) | 3 | 2
Abdominal tenderness (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haematochezia (Gastrointestinal disorders) | 3 | 0
Retching (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Abdominal rigidity (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 25 | 15
Disease progression (General disorders) | 1 | 2
Pyrexia (General disorders) | 23 | 9
Asthenia (General disorders) | 9 | 6
Oedema peripheral (General disorders) | 8 | 9
Pain (General disorders) | 8 | 6
Chills (General disorders) | 9 | 5
Chest pain (General disorders) | 4 | 1
Gait disturbance (General disorders) | 3 | 1
Malaise (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 2 | 2
Hepatomegaly (Hepatobiliary disorders) | 3 | 0
Urinary tract infection (Infections and infestations) | 6 | 1
Pneumonia (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 11 | 4
Incision site pain (Injury, poisoning and procedural complications) | 6 | 8
Incision site complication (Injury, poisoning and procedural complications) | 4 | 1
Gamma-glutamyltransferase increased (Investigations) | 18 | 7
Blood alkaline phosphatase increased (Investigations) | 16 | 7
Haemoglobin decreased (Investigations) | 13 | 8
Weight decreased (Investigations) | 13 | 8
Blood albumin decreased (Investigations) | 14 | 6
Blood calcium decreased (Investigations) | 9 | 6
Blood glucose increased (Investigations) | 9 | 3
Aspratate aminotransferase increased (Investigations) | 6 | 3
Blood sodium increased (Investigations) | 6 | 3
Alanine aminotransferase increased (Investigations) | 2 | 4
Blood bilirubin increased (Investigations) | 5 | 1
Body temperature increased (Investigations) | 4 | 2
Blood creatinine increased (Investigations) | 5 | 0
Blood potassium increased (Investigations) | 2 | 2
Blood pressure increased (Investigations) | 3 | 1
Lipase increased (Investigations) | 3 | 0
Weight increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 17 | 6
Anorexia (Metabolism and nutrition disorders) | 12 | 9
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 5 | 2
Hypoaethesia (Nervous system disorders) | 4 | 0
Neuropathy (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 0 | 2
Speech disorder (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 5 | 9
Depression (Psychiatric disorders) | 7 | 6
Insomnia (Psychiatric disorders) | 8 | 5
Confusional state (Psychiatric disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 2 | 4
Pollakiuria (Renal and urinary disorders) | 3 | 3
Chromaturia (Renal and urinary disorders) | 2 | 1
Micturition urgency (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 7
Rash (Skin and subcutaneous tissue disorders) | 9 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hot flush (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 3 | 0
Lymphoedema (Vascular disorders) | 2 | 1
Flushing (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Limitations of this study include the lack of non-macrobead implanted comparator groups for pancreatic and mCRC subjects, the small sample sizes of both groups, the limited number of subjects with >1 implant and the potential for various biases due to the non-randomized study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor retains the first right for scientific disclosure of study results. PI may draft a study results disclosure for scientific publication following the earlier of sponsor's disclosure or 12 months after study completion at all sites. Sponsor has 60 days to review PI's draft for patentable subject matter or confidential information. PI will delete any confidential information and delay any disclosure for another 60 days for sponsor to secure proprietary protection.

DOCUMENTS (3):
  • Study Protocol (2014-11-12): https://cdn.clinicaltrials.gov/large-docs/13/NCT01053013/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT01053013/SAP_001.pdf
  • Informed Consent Form (2015-03-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT01053013/ICF_002.pdf